CLINICAL TRIAL: NCT01823198
Title: NK Cells With HLA Compatible Hematopoietic Transplantation for High Risk Myeloid Malignancies
Brief Title: Donor Natural Killer Cells and Donor Stem Cell Transplant in Treating Patients With High Risk Myeloid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0819; NCI-2013-00993 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RP110553-P3; 2012-0819 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Erythroid Leukemia; Acute Megakaryoblastic Leukemia; Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Acute Myeloid Leukemia in Remission; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Blasts Under 20 Percent of Bone Marrow Nucleated Cells; Blasts Under 20 Percent of Peripheral Blood White Cells; Chronic Myelomonocytic Leukemia; High Risk Myelodysplastic Syndrome; Myelodysplastic Syndrome; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Therapy-Related Acute Myeloid Leukemia; Therapy-Related Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Acute; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — aldesleukin; Busulfan; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (NK cells, PBSC transplant) (Experimental): Patients receive fludarabine phosphate IV over 1 hour and busulfan IV over 3 hours on days -13 to -10. Patients then receive allogeneic CD56-positive CD3-negative natural killer cells IV over 1 hour on day -8. Patients also receive aldesleukin SC QD on days -8 to -4. Patients then undergo allogeneic PBSC transplant on day 0.
  Interventions: Biological: Aldesleukin; Biological: Allogeneic CD56-positive CD3-negative Natural Killer Cells; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Allogeneic CD56-positive CD3-negative Natural Killer Cells — Given IV
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic PBSC transplant
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSC transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of donor natural killer cells when given together with donor stem cell transplant and to see how well they work in treating patients with myeloid malignancies that are likely to come back or spread. Giving chemotherapy, such as busulfan and fludarabine phosphate, before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells and natural killer cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety of infusing ex vivo expanded natural killer (NK) cells in patients receiving busulfan-fludarabine phosphate (fludarabine) with an allogeneic human leukocyte antigen (HLA) matched hematopoietic transplantation for myeloid malignancies. Two sources of NK cells could be studied, depending on what donor source is available: cells from the HLA matched related donor or cells from an unrelated cord blood unit.

II. For each source of NK cells: the maximum tolerated cell dose; the phenotype and function of the ex vivo expanded NK cells and their survival in vivo; the rate of engraftment, graft-vs.-host disease (GVHD), immune reconstitution, relapse rates and survival for patients receiving this regimen will be determined.

OUTLINE: This is a phase I, dose-escalation study of NK cells followed by a phase II study.

Patients receive fludarabine phosphate intravenously (IV) over 1 hour and busulfan IV over 3 hours on days -13 to -10. Patients then receive allogeneic CD56-positive CD3-negative natural killer cells IV over 1 hour on day -8. Patients also receive aldesleukin subcutaneously (SC) once daily (QD) on days -8 to -4. Patients then undergo allogeneic peripheral blood stem cell (PBSC) transplant on day 0.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia who fail to achieve complete remission with one course of induction chemotherapy or after relapse; patients must have less than 20% bone marrow or peripheral blood blasts
* Acute myeloid leukemia in first remission with any of the following high risk features defined as:

  * Adverse cytogenetics: -5, deletion (del) 5q, -7, del7q, abnormalities involving 3q, 9q, 11q, 20q, 21q, 17, +8 or complex karyotype (> 3 abnormalities)
  * Preceding myelodysplastic or myeloproliferative syndrome
  * Presence of high risk molecular abnormalities including FLT3 mutations, DNMT3A, TET2; ras; kit
  * French-American-British (FAB) monosomy (M)6 or M7 classification
  * Treatment related acute myeloid leukemia (AML)
  * Residual cytogenetic or molecular abnormalities
* Myelodysplastic syndromes with intermediate, high or very high risk Revised International Prognostic Scoring System (R-IPSS) score, chronic myelomonocytic leukemia (CMML) or therapy related myelodysplastic syndromes (MDS)
* Chronic myeloid leukemia (CML) which:

  * Failed to achieve a cytogenetic remission to tyrosine kinase inhibitor treatment or has a cytogenetic relapse
  * Has ever been in accelerated phase or blast crisis
* Patient must have an identified HLA (A,B,C,DR) compatible related or unrelated donor who is age 16 years of age or older and weighs at least 110 pounds for the stem cell donation
* Zubrod performance status 0 to 2 or Karnofsky of at least 60
* Left ventricular ejection fraction >= 45%; no uncontrolled arrhythmias or uncontrolled symptomatic cardiac disease
* Forced expiratory volume in one second (FEV1) >= 50% of expected, corrected for hemoglobin
* Forced vital capacity (FVC) >= 50% of expected, corrected for hemoglobin
* Diffusing capacity of the lung for carbon monoxide (DLCO) >= 50% of expected, corrected for hemoglobin
* Bilirubin =< 1.5 mg/dl (unless Gilbert's syndrome)
* Serum glutamate pyruvate transaminase (SGPT) =< 200 IU/ml unless related to patient malignancy
* Hepatitis B surface antigen negative and hepatitis C antibody negative
* No evidence of chronic active hepatitis or cirrhosis
* Patients with a history of hepatitis C, but have a negative viral load, are eligible
* The protocol chairman will determine the eligibility of patients related to hepatic abnormalities
* Serum creatinine < 1.5 mg%
* Patient or patient's legal representative, parent(s) or guardian able to sign informed consent; patients aged 7 to < 18 to provide assent
* Pediatric patients (age 7-18 years) will be entered only after 3 adult patients have been entered without dose limiting toxicity

Exclusion Criteria:

* Uncontrolled infection, not responding to appropriate antimicrobial agents after seven days of therapy; the protocol principal investigator (PI) is the final arbiter of eligibility
* Pleural/pericardial effusion or ascites > 1 L
* Patients who are known to be human immunodeficiency virus (HIV)-seropositive
* Pregnancy: positive pregnancy test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization
* Women of child bearing potential not willing to use an effective contraceptive measure while on study
* Patients who are known to have allergy to mouse proteins

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Champlin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at MD Anderson Cancer Center.
Pre-assignment Details: Sixty three participants were enrolled in MDACC which 42 recipients and 21 related donors have signed consents. Twenty one ex-vivo NK cell derived from cord blood are from MDACC cord blood bank.
Groups:
- Phase I: NK Cell Dose Level 1_10^6; Phase I: NK Cell Dose Level 2_10^7; Phase I: NK Cell Dose Level 3_ 3x10^7: Allogeneic stem cell transplant for patients with high risk myeloid malignancies conditioned with Fludarabine and Busulfan in combination with ex vivo expanded NK cells from 3 different NK cell sources : KIR mismatched haplo donors, KIR mismatched cord blood donors or HLA matched related donors.
- Phase I: NK Cell Dose Level 4_ 10^8; Phase II: NK Cell Dose Level 4_ 10^8: Allogeneic stem cell transplant for patients with high risk myeloid malignancies conditioned with Fludarabine and Busulfan in combination with phase I/II escalation ex vivo expanded NK cells from 3 different NK cell sources : KIR mismatched haplo donors, KIR mismatched cord blood
- Phase II: NK Cell Dose Level 3_3x10^7: Allogeneic stem cell transplant for patients with high risk myeloid malignancies conditioned with Fludarabine and Busulfan in combination with phase I/II escalation ex vivo expanded NK cells from 3 different NK cell sources : KIR mismatched haplo donors, KIR mismatched cord blood donors or HLA matched related donors.
- Donors: Donors: KIR mismatched haplo donors, KIR mismatched cord blood donors or HLA matched related donors.
Period: Overall Study
Arm/Group | Phase I: NK Cell Dose Level 1_10^6 | Phase I: NK Cell Dose Level 2_10^7 | Phase I: NK Cell Dose Level 3_ 3x10^7 | Phase I: NK Cell Dose Level 4_ 10^8 | Phase II: NK Cell Dose Level 3_3x10^7 | Phase II: NK Cell Dose Level 4_ 10^8 | Donors
Started | 6 | 6 | 4 | 4 | 1 | 21 | 21
Completed | 6 | 5 | 4 | 4 | 1 | 18 | 18
Not Completed | 0 | 1 | 0 | 0 | 0 | 3 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Donor participants only signed the consents and were not part of the results and Adverse events were not collected.
Groups:
- Phase I: NK Cell Dose Level 4_ 10^8; Phase II: NK Cell Dose Level 3_3x10^7: Allogeneic stem cell transplant for patients with high risk myeloid malignancies conditioned with Fludarabine and Busulfan in combination with phase I/II escalation ex vivo expanded NK cells from 3 different NK cell sources : KIR mismatched haplo donors, KIR mismatched cord blood donors or HLA matched related donors.
- Total: Total of all reporting groups
Arm/Group | Phase I: NK Cell Dose Level 1_10^6 | Phase I: NK Cell Dose Level 2_10^7 | Phase I: NK Cell Dose Level 3_ 3x10^7 | Phase I: NK Cell Dose Level 4_ 10^8 | Phase II: NK Cell Dose Level 3_3x10^7 | Phase II: NK Cell Dose Level 4_ 10^8 | Donors | Total
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 1 | 21 | 21 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Between 18 and 65 years | 6 | 6 | 4 | 4 | 1 | 20 | 21 | 62
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 2 | 0 | 5 | 12 | 28
  Male | 3 | 3 | 1 | 2 | 1 | 16 | 9 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 0 | 1 | 0 | 4 | 6 | 16
  Not Hispanic or Latino | 3 | 4 | 4 | 3 | 1 | 17 | 15 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 4 | 4 | 1 | 21 | 21 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-limiting Toxicities (DLT)
Description: Participants that experienced DLT related to the NK Cells post transplant at different dose levels.
Time Frame: Up to 42 days
Population: Twenty one donor participants were not included in outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: NK Cell Dose Level 1_10^6 | Phase I: NK Cell Dose Level 2_10^7 | Phase I: NK Cell Dose Level 3_ 3x10^7 | Phase I: NK Cell Dose Level 4_ 10^8 | Phase II: NK Cell Dose Level 3_3x10^7 | Phase II: NK Cell Dose Level 4_ 10^8
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 1 | 21
Participants
  Group A: NK cells from KIR mismatched haplo donors | 2 | 1 | 0 | 0 | 0 | 0
  Group B: NK cells from KIR mismatched cord blood donors | 2 | 2 | 2 | 2 | 1 | 12
  Group C: NK cells from matched related donors | 2 | 3 | 2 | 2 | 0 | 9

2. Secondary Outcome: Overall Survival
Description: Participants that survived between day of transplant and day of death on different dose levels.
Time Frame: Up to 2 years
Population: Twenty one donor participants were not included in outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: NK Cell Dose Level 1_10^6 | Phase I: NK Cell Dose Level 2_10^7 | Phase I: NK Cell Dose Level 3_ 3x10^7 | Phase I: NK Cell Dose Level 4_ 10^8 | Phase II: NK Cell Dose Level 3_3x10^7 | Phase II: NK Cell Dose Level 4_ 10^8
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 1 | 21
Participants
  Group A: NK cells from KIR mismatched haplo donors | 2 | 0 | 0 | 0 | 0 | 0
  Group B: NK cells from KIR mismatched cord blood donors | 1 | 1 | 0 | 1 | 1 | 7
  Group C: NK cells from matched related donors | 2 | 0 | 3 | 2 | 0 | 2

3. Secondary Outcome: Number of Participants With Grade 3 Toxicities
Description: Number of participants that had grade 3 toxicities up to day 42.
Time Frame: Up to day 42
Population: Twenty one donor participants were not included in outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: NK Cell Dose Level 1_10^6 | Phase I: NK Cell Dose Level 2_10^7 | Phase I: NK Cell Dose Level 3_ 3x10^7 | Phase I: NK Cell Dose Level 4_ 10^8 | Phase II: NK Cell Dose Level 3_3x10^7 | Phase II: NK Cell Dose Level 4_ 10^8
Number analyzed (Participants) | 6 | 6 | 4 | 4 | 1 | 21
Participants
  Group A: NK cells from KIR mismatched haplo donors | 2 | 1 | 0 | 0 | 0 | 0
  Group B: NK cells from KIR mismatched cord blood donors | 1 | 2 | 1 | 1 | 1 | 11
  Group C: NK cells from matched related donors | 2 | 2 | 2 | 2 | 0 | 6

ADVERSE EVENTS:
Time Frame: Up to 42 days. All-Cause Mortality was monitored/assessed for up to 2 years).
Description: Donor participants only signed the consents and were not part of the results and Adverse events were not collected.
Arm/Group | Phase I: NK Cell Dose Level 1_10^6 | Phase I: NK Cell Dose Level 2_10^7 | Phase I: NK Cell Dose Level 3_ 3x10^7 | Phase I: NK Cell Dose Level 4_ 10^8 | Phase II: NK Cell Dose Level 3_3x10^7 | Phase II: NK Cell Dose Level 4_ 10^8 | Donors
All-Cause Mortality (participants affected / at risk) | 1/6 | 4/6 | 2/4 | 1/4 | 0/1 | 9/21 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 1/4 | 0/4 | 1/1 | 6/21 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 4/4 | 4/4 | 1/1 | 17/21 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: NK Cell Dose Level 1_10^6 (N=6) | Phase I: NK Cell Dose Level 2_10^7 (N=6) | Phase I: NK Cell Dose Level 3_ 3x10^7 (N=4) | Phase I: NK Cell Dose Level 4_ 10^8 (N=4) | Phase II: NK Cell Dose Level 3_3x10^7 (N=1) | Phase II: NK Cell Dose Level 4_ 10^8 (N=21) | Donors (N=0)
Viral Infections (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic lung GvHD (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Secondary graft failure (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal Infections (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver GvHD (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
GI GvHD (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic Skin GvHD (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver GvHD (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Bacterial Infections (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: NK Cell Dose Level 1_10^6 (N=6) | Phase I: NK Cell Dose Level 2_10^7 (N=6) | Phase I: NK Cell Dose Level 3_ 3x10^7 (N=4) | Phase I: NK Cell Dose Level 4_ 10^8 (N=4) | Phase II: NK Cell Dose Level 3_3x10^7 (N=1) | Phase II: NK Cell Dose Level 4_ 10^8 (N=21) | Donors (N=0)
ABO incompatibility (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bacterial Infections (Infections and infestations) | 2 | 0 | 2 | 2 | 1 | 7 | 0
BK virus associated hemorrhagic cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 5 | 0
Bronchiolitis obliterans with organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic Liver GvHD (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic ocular GvHD (Eye disorders) | 2 | 1 | 1 | 1 | 0 | 7 | 0
Chronic oral GvHD (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 6 | 0
Chronic Skin GvHD (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 0 | 1 | 0
Chronic vaginal GvHD (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 0 | 3 | 0 | 10 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Ejection fraction decreased (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Elevated bilirubin (Investigations) | 1 | 3 | 0 | 1 | 1 | 8 | 0
Elevated transminitis (Investigations) | 2 | 1 | 0 | 1 | 0 | 6 | 0
Fevers (General disorders) | 0 | 3 | 2 | 3 | 0 | 4 | 0
Flu like syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fluid overload (General disorders) | 4 | 2 | 3 | 1 | 0 | 9 | 0
Fungal Infections (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
GI GvHD (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 5 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 3 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 0 | 3 | 0
Idiopathic thrombocytopenic purpura (ITP) (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver GvHD (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Mucositis (Gastrointestinal disorders) | 6 | 5 | 4 | 4 | 1 | 17 | 0
Nausea (Gastrointestinal disorders) | 6 | 5 | 3 | 4 | 1 | 17 | 0
Neutropenic fevers (Blood and lymphatic system disorders) | 3 | 2 | 2 | 1 | 0 | 7 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 1 | 5 | 0
Skin GvHD (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 2 | 1 | 10 | 0
Upper GI GvHD (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 4 | 0
Viral Infections (Infections and infestations) | 4 | 2 | 2 | 2 | 1 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT01823198/Prot_SAP_000.pdf